CLINICAL TRIAL: NCT04353856
Title: Evolution of the Quality of Life During a Twin Pregnancy
Brief Title: Quality of Life During a Twin Pregnancy
Acronym: QUALIGEM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0138; ID-RCB (Other: 2020-A00385-34)
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Twin Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- twin pregnancy: Women followed for a twin pregnancy
  Interventions: Other: quality of life assessment

INTERVENTIONS:
Other: quality of life assessment — quality of life assessment using the EQ5D questionnaire once a month

SUMMARY:
Quality of life has recently appeared as a component of health. Pregnancy has an impact on the quality of life of the parturient, whether through physical or psychological changes.

It is common to think that quality of life is altered in the context of a twin pregnancy, but this has never been scientifically demonstrated.

The hypothesis is to observe a decrease in the quality of life of pregnant women with twins at the end of pregnancy, in particular in case of a pregnancy-related pathology.

ELIGIBILITY:
Inclusion Criteria:

* woman over 18
* ongoing twin pregnancy (2 live fetuses)
* pregnancy <15 weeks (weeks of gestation) completed
* patient with follow-up at the Hôpital Femme Mère Enfant
* person having expressed her non-opposition

Exclusion Criteria:

* inability to understand the information given and the questionnaire
* person deprived of liberty, under guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women over 18 years old, followed for a twin pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Quality of life EQ5D questionnaire | Month 3
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L).
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Quality of life EQ5D questionnaire | Month 4
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L)
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Quality of life EQ5D questionnaire | Month 5
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L)
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Quality of life EQ5D questionnaire | Month 6
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L)
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Quality of life EQ5D questionnaire | Month 7
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L)
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Quality of life EQ5D questionnaire | Month 8
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L)
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Quality of life EQ5D questionnaire | Month 9
  Quality of life score established by the EQ5D questionnaire (EUROQOL EQ-5D-3L)
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No